CLINICAL TRIAL: NCT04474301
Title: Well-Being and Quality of Life in Melanoma Patients During COVID-19 Pandemic
Brief Title: Well-Being and Health-Related Quality of Life in Melanoma Patients During COVID-19 Pandemic
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2020-0470; NCI-2020-04587 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0470 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-07-14; First posted 2020-07-16 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: COVID-19 Infection; Melanoma
MeSH Terms: conditions — COVID-19; Melanoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (survey administration): Patients complete a survey over 10 minutes.
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Survey Administration — Complete survey

SUMMARY:
The primary purpose of this study is to gain an understanding of how experiences during the COVID-19 pandemic, regardless of COVID-19 status, may have impacted multiple domains of health-related quality of life and other areas such as COVID-19 specific psychological distress, and disruptions to health care, finances and social interactions. We will also evaluate the extent to which resiliency factors such as social support, perceived benefits under times of stress, and ability to manage stress may buffer associations between COVID-19 experiences and HRQoL. To meet these objectives, we have developed a 10-minute questionnaire that taps into these areas and is based on prior work addressing concerns of other pandemics or national crises. Participants will have previously consented to protocol PA15-0336 and have provided prior lifestyle data. This will allow us to connect the COVID-19 survey data with prior existing data.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess experiences during the COVID-19 pandemic (e.g., exposure, risk factors, testing, isolation, seropositivity, hospitalization, loss of family or friends); COVID-19-specific psychological distress (e.g., fear, anxiety and depressive symptoms); health, financial and social disruptions; perceived benefits and social support; and health-related quality of life (HRQoL) in melanoma patients who participated in protocol PA15-0336.

II. Evaluate the extent to which COVID-19 experiences are associated with COVID-19-specific psychological distress, health, financial and social disruptions, perceived benefits and social support, and HRQoL.

III. Evaluate the extent to which resiliency factors such as social support and perceived benefits moderate the effects of COVID-19 experiences on COVID-19-specific psychological distress and HRQoL.

IV. Explore the association between prior lifestyle data collected as part of PA15-0336 and COVID-19-specific psychological distress and HRQoL.

OUTLINE:

Patients complete a survey over 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have signed consent for PA15-0336
* Has an active email address and can be contacted via MyChart
* Documentation of being alive per the cancer registry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have signed consent for PA15-0336.
Sampling Method: Non-Probability Sample
Enrollment: 1152 (Estimated)
Dates: Start 2020-06-11 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Experiences during the COVID-19 pandemic | Survey completion Up to 2 months
  Including exposure, risk factors, testing, isolation, seropositivity, hospitalization, or loss of family or friends.
COVID-19-specific psychological distress | Survey completion Up to 2 months
COVID-19-specific health | Survey completion Up to 2 months
COVID-19-specific financial and social disruptions | Survey completion Up to 2 months
COVID-19-specific perceived benefits and social support | Survey completion Up to 2 months
COVID-19-specific health related quality of life (HRQoL) | Survey completion Up to 2 months
Effects of COVID-19 experiences on COVID-19-specific psychological distress and HRQoL | Survey completion Up to 2 months
  Will evaluate the extent to which resiliency factors such as social support and perceived benefits moderate the effects of COVID-19 experiences on COVID-19-specific psychological distress and HRQoL.
Prior lifestyle data | Survey completion Up to 2 months
  Will explore the association between prior lifestyle data collected as part of PA15-0336 and COVID-19-specific psychological distress and HRQoL.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Cohen, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org